CLINICAL TRIAL: NCT00020111
Title: Phase I Trial and Pharmacokinetic Study of Arsenic Trioxide in Pediatric Patients With Refractory Leukemia or Lymphoma
Brief Title: Arsenic Trioxide in Treating Young Patients With Refractory Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067717; NCI-00-C-0070J; NCI-T99-0080; NCT00004548 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2005-02

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent childhood acute myeloid leukemia; childhood acute promyelocytic leukemia (M3); recurrent childhood acute lymphoblastic leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma; childhood chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of arsenic trioxide in treating young patients with leukemia or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of arsenic trioxide in pediatric patients with refractory leukemia or lymphoma.
* Determine the maximum tolerated dose of this drug in this patient population.
* Determine the plasma pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to disease (acute promyelocytic leukemia [APL] vs non-APL).

* Stratum I (APL patients): Patients receive standard-dose arsenic trioxide IV over 2 hours daily 5 days a week for 4 weeks. Treatment continues every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
* Stratum II (Non-APL patients): Cohorts of 3-6 patients receive escalating doses of arsenic trioxide (according to the stratum 1 schedule above) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive treatment with arsenic trioxide at the recommended phase II dose.

Leukemia patients in both strata without progressive disease who have not achieved complete remission after the first 20 doses may continue to receive arsenic trioxide for 2 additional weeks.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A maximum of 18 patients will be accrued for stratum I of this study within 2-3 years. A total of 3-30 patients will be accrued for stratum II of this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed leukemia or lymphoma refractory to standard curative treatment regimens
* Measurable or evaluable disease
* No meningeal leukemia or lymphoma
* No HIV-related lymphoma
* No lymphoproliferative diseases

PATIENT CHARACTERISTICS:

Age:

* 2 to 21

  * Acute promyelocytic leukemia (APL) patients (stratum I) must be age 2 to 12

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin normal
* SGPT less than 2 times upper limit of normal
* No significant hepatic dysfunction that would preclude study therapy

Renal:

* Creatinine normal (age adjusted) OR
* Creatinine clearance at least 60 mL/min
* Potassium, magnesium, and calcium at least lower limit of normal (oral or IV supplementation allowed)
* No significant renal dysfunction that would preclude study therapy

Cardiovascular:

* Rate corrected QTc interval no greater than 0.48 on EKG
* No significant cardiac dysfunction that would preclude study therapy
* No cardiac disease, including dysrhythmias

Pulmonary:

* No significant pulmonary dysfunction that would preclude study therapy

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No persistent grade 3 or greater sensory or motor neuropathy
* No prior grand mal seizures (grade 3 or greater) within the past 2 years other than febrile seizures (except for patients with APL at discretion of investigator)
* No clinically significant unrelated systemic illness that would preclude study therapy (e.g., serious infection)
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior colony-stimulating factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF], and epoetin alfa)
* No concurrent immunotherapy

Chemotherapy:

* No prior arsenic trioxide
* At least 2 weeks since prior chemotherapy (4 weeks for nitrosoureas) and recovered
* No concurrent intrathecal chemotherapy except for acute promyelocytic leukemia (APL) patients experiencing progressive meningeal leukemia and demonstrating benefit from arsenic trioxide for systemic disease
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No concurrent steroids (except corticosteroids for retinoic acid syndrome)

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* At least 6 months since prior anticonvulsants
* At least 1 week since prior retinoid therapy
* No concurrent retinoids
* No other concurrent investigational agents

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Frank M. Balis, MD, Study Chair — National Cancer Institute (NCI)
Locations (52):
- United States (47):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - County of Los Angeles Harbor-UCLA Medical Center, Torrance, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Simmons Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Fox E, Razzouk BI, Widemann BC, Xiao S, O'Brien M, Goodspeed W, Reaman GH, Blaney SM, Murgo AJ, Balis FM, Adamson PC. Phase 1 trial and pharmacokinetic study of arsenic trioxide in children and adolescents with refractory or relapsed acute leukemia, including acute promyelocytic leukemia or lymphoma. Blood. 2008 Jan 15;111(2):566-73. doi: 10.1182/blood-2007-08-107839. Epub 2007 Oct 24. PMID 17959855
- [Result] Fox E, Adamson PC, Murgo A, et al.: Phase 1 trial and pharmacokinetic study of arsenic trioxide in children with refractory leukemia. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1582, 2002.